CLINICAL TRIAL: NCT01005732
Title: Effectiveness of Pressure Garment Therapy After Burns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Dr. Loren Engrav, University of Washington
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 30336-B; H133G050022; NIDRR_UWashingtonBMS_pgarment
Record Dates: First submitted 2009-10-30; First posted 2009-11-02 (Estimated); Results first posted 2011-04-04 (Estimated); Last update posted 2011-04-04 (Estimated); Status verified 2011-04

CONDITIONS: Hypertrophic Scarring After Burn Injury
Keywords: hypertrophic; scar; burn; cicatrix; pressure; garment
MeSH Terms: conditions — Hypertrophy; Cicatrix; Burns

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Custom fabricated pressure garments — Cloth garments designed to apply 17-24 mmHg pressure to the 1/2 the burn wound and <5 mmHg to the other half, to be worn 23 hours per day until wounds mature, approximately 12 months
  Other Names: Medical Z (Medical Z, San Antonio, TX)

SUMMARY:
Purpose - To determine the effectiveness of custom-fit pressure garment therapy in the prevention of hypertrophic scarring in healed burns.

Background - Approximately one million people are burned each year in the United States. The most devastating outcomes following burns is the ugly, itchy, hypertrophic scar that interferes with work and all other aspects of life. Pressure garment therapy is routinely used to minimize hypertrophic scarring even though there is no scientifically valid data that this therapy is efficacious. Pressure garments are extremely unattractive, expensive and uncomfortable and their use needs to be based upon valid data.

Goals and Objectives - The investigators plan to determine the effectiveness of pressure garment therapy in the control of hypertrophic scarring in healed burns.

Methods - The I-Scan® device was designed to measure pressure at the body/environment interface and allows clinicians to deal with pressure-related problems for at-risk patients. It has been widely used in rehabilitation medicine but not with burn survivors. The investigators will use this device to measure the pressure at the garment/skin interface. 2) Furthermore, the few studies that have been attempted to determine efficacy have used between subjects designs. Since burn depth is extremely variable from patient to patient and since hypertrophic scarring is greatly influenced by age and race/origin, the between subjects design requires very large numbers of subjects. The investigators will use a within wounds design studying forearm burns and applying pressure to half of the wound and no pressure to the other half. The investigators will then compare hardness, color, thickness and clinical appearance.

ELIGIBILITY:
Inclusion Criteria:

* Treated from time of burn at the University of Washington Burn Center during the first two years of the grant period
* Burns covering the majority of the forearm that healed spontaneously in three or more weeks. Patients will be entered into the study within 4 weeks of injury.
* Age 7-65 years. Patients younger than 7 years will be excluded given the cooperation required during follow-up evaluations. Patients over 65 years will be excluded since the incidence of hypertrophic scarring in persons over 65 is too low to warrant pressure garment trials.
* Patients of any race, ethnicity, or skin color.
* Informed, written consent in accord with the rules of the Human Subjects Committee of the University of Washington and the Health Insurance Portability and Accountability Act (HIPAA).

Exclusion Criteria:

* Incarcerated patients
* Homeless patients
* Patients with substance abuse
* Patients with psychiatric diagnosis
* Patients unavailable to return regularly for follow-up evaluations

Ages: 7 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 1995-11; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Loren Engrav, Principal Investigator — University of Washington
Locations (1):
- University of Washington Burn Center, Seattle, Washington, United States

REFERENCES:
- [Background] Engrav LH, Heimbach DM, Rivara FP, Moore ML, Wang J, Carrougher GJ, Costa B, Numhom S, Calderon J, Gibran NS. 12-Year within-wound study of the effectiveness of custom pressure garment therapy. Burns. 2010 Nov;36(7):975-83. doi: 10.1016/j.burns.2010.04.014. Epub 2010 Jul 1. PMID 20537469

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During the 12-year period from 1995 to 2007, in accord with the Human Subjects Division of the University of Washington, 67 consecutive patients were enrolled. Thirteen patients exited the study prior to any data collection. Eleven of these chose to remove themselves, one was lost to follow-up and the reason was not recorded for one patient.
Groups:
- Pressure Garment on Burn Wound: Pressure garment therapy was started within 2 weeks of re-epithelialization. A custom-fit pressure garment was fabricated by Medical Z Inc. (Medical Z, San Antonio, TX) and designed such that it applied pressure to only one-half of the wound, proximal or distal (according to coin toss by a consistent individual not involved in data collection for the study). The standard Lycra® 6-way stretch fabric was designed to apply 17-24 mm Hg to the normal/high compression zone and <5 mm Hg to the low compression zone. Subjects were instructed to wear the garments 23 hours per day, removing them only for bathing.
Period: Overall Study
Arm/Group | Pressure Garment on Burn Wound
Started | 54
Completed | 43
Not Completed | 11
Not completed — Lost to Follow-up | 10
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pressure Garment on Burn Wound
Number analyzed (Participants) | 54
Age Continuous [Mean (Standard Deviation); unit: years] | 36 (14)
Age, Customized [Number; unit: participants]
  7-14 years | 3
  15-30 years | 17
  31-59 years | 34
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 46
Region of Enrollment [Number; unit: participants]
  United States | 54

OUTCOME MEASURES:

1. Primary Outcome: Pressure Under Compression Garment
Description: Pressure measurements were obtained at the scar/garment interface using the I-ScanTM System (Tekscan, Inc., South Boston, MA). The device was calibrated and the pressure determined in mmHg. Pressure measurements were obtained by a therapist not involved in the care of the patient, who was trained in the use of the device. Therefore pressure ''dose'' was measured directly. Values reported are averaged over indicated visits.
Time Frame: Approximately 2.5, 5, 7.5, 10, and 12 months (follow-up visits 1-5)
Population: All Participants with available and evaluable measurement.
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Normal/High Pressure Zone: Normal/high compression area of custom-fit compression garment applied to 1/2 of patient's wound (randomly assigned to proximal/distal)
- Low Compression Zone: Low compression area of custom-fit compression garment applied to 1/2 of patient's wound (randomly assigned to proximal/distal)
Arm/Group | Normal/High Pressure Zone | Low Compression Zone
Number analyzed (Participants) | 50 | 50
mm Hg | 25 (6.3) | 6.4 (6.2)

2. Secondary Outcome: Durometer (Hardness) of Wound
Description: A single Rex Durometer Hand Model 1600, Type 00, without a foot attachment (Rex Gauge Company Inc., Glenview, IL) was used to measure scar hardness throughout the study. This device measures hardness of light foams, sponge rubber gels, and animal tissue in "durometer units" (range 0=soft, 100=hard). Measurements were obtained with the person in the sitting position with the forearm supported in a horizontal position on a desk and the shoulder adducted. The area of interest was triangulated and measurements obtained at the corners were averaged; the sides of the triangle were 3-5 cm.
Time Frame: Approximately 2.5, 5, 7.5, 10, and 12 months (follow-up visits 1-5)
Population: All Participants with available and evaluable measurement.
Measure: Mean (Standard Deviation); unit: durometer units
Groups:
- Kneecap: Hardness of uninjured skin over a bony prominence is provided for comparison.
- Uninjured Forearm Skin: Hardness of uninjured forearm skin is provided for comparison.
Arm/Group | Normal/High Pressure Zone | Low Compression Zone | Kneecap | Uninjured Forearm Skin
Number analyzed (Participants) | 54 | 54 | 54 | 54
durometer units
  Study Period 1 (n=51) | 47 (7) | 46 (6) | 72 (9) | 39 (4)
  Study Period 2 (n=44) | 46 (8) | 49 (7) | NA (NA) — Measurement made at only one visit. | NA (NA) — Measurement made at only one visit.
  Study Period 3 (n=37) | 47 (7) | 48 (8) | NA (NA) — Measurement made at only one visit. | NA (NA) — Measurement made at only one visit.
  Study Period 4 (n=33) | 45 (7) | 48 (7) | NA (NA) — Measurement made at only one visit. | NA (NA) — Measurement made at only one visit.
  Study Period 5 (n=26) | 45 (7) | 49 (7) | NA (NA) — Measurement made at only one visit. | NA (NA) — Measurement made at only one visit.

3. Secondary Outcome: Color of Wound
Description: A Chromameter Minolta CR-300 (Konica Minolta, Ramsey, NJ) measured skin color. Skin surface illuminated by pulsed xenon arc lamp. Light reflected perpendicular to surface collected for a tri-stimulus color analysis. One measurement consisted of three flashes of illumination in order to obtain a mean value. Measurement values are in the L*a*b* color space was described by The Commission Internationale de I'Eclairage (CIE)(L=brightness [100=white,0=black], a=red-green[red=60,green=-60], b=yellow-blue[yellow=60,blue=-60])
Time Frame: Approximately12 months (follow-up visits 5)
Population: All Participants with available and evaluable measurement.
Measure: Mean (Standard Deviation); unit: color space parameter units
Units Other Than Participants: Colorimeter observations
Arm/Group | Normal/High Pressure Zone | Low Compression Zone
Number analyzed (Participants) | 31 | 31
Number analyzed (Colorimeter observations) | 81 | 81
color space parameter units
  L color parameter | 56.3 (18.6) | 55.2 (17.6)
  a color parameter | 9 (9.7) | 9.5 (9.2)
  b color parameter | 8.2 (3.2) | 8.5 (3.2)

4. Secondary Outcome: Thickness of Wound
Description: Scar thickness in millimeters was obtained with high-frequency ultrasonography in the Department of Radiology. Several machines and probes were used over the years each with accuracy to 0.5 mm. The area of interest was triangulated and measurements obtained at the corners were averaged; the sides of the triangle were 3-5 cm.
Time Frame: Approximately 12 months (follow-up visit 5)
Population: All Participants with available and evaluable measurement.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Normal/High Pressure Zone | Low Compression Zone
Number analyzed (Participants) | 28 | 28
mm | 2.8 (3.2) | 3.4 (3.0)

5. Secondary Outcome: Clinical Appearance of Wound
Description: Photographs of wounds showed final cosmetic result. The two compression areas for each photograph were labeled distal (D) and proximal (P). We asked 11 experts (blinded as to the compression of the rated zones) to judge which zone (D or P) had the better cosmetic appearance or whether there was no difference. Votes were tallied according to the unblinded compression zone (i.e., high/normal and low). We report number of participants for which the rating experts all agreed or did not all agree (i.e., voted the other zone or "no difference") that the indicated zone had the better appearance.
Time Frame: Approximately 12 months (follow-up visit 5)
Population: All Participants with available and evaluable measurement.
Measure: Number; unit: Participants
Arm/Group | Normal/High Pressure Zone | Low Compression Zone
Number analyzed (Participants) | 28 | 28
Participants
  All experts agree zone has better appearance | 3 | 0
  All experts do not agree zone has better appearanc | 38 | 41

6. Secondary Outcome: Compliance With Wearing Compression Garment
Description: The patients were asked to complete a compliance form indicating how many hours the garment was worn each day.
Time Frame: About 12 months (follow-up visit 5)
Population: All Participants with available and evaluable data.
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | Pressure Garment on Burn Wound
Number analyzed (Participants) | 27
hours per day | 20.4 (3.9)

ADVERSE EVENTS:
Arm/Group | Pressure Garment on Burn Wound
Serious Adverse Events (participants affected / at risk) | 0/54
Other Adverse Events (participants affected / at risk) | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No